CLINICAL TRIAL: NCT06800586
Title: Tumors and Respiratory System Diseases Due to Air Pollution: New Biomarkers of Exposure and Effects
Acronym: RECAP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RECAP; PNRR-MCNT1-2023-12378402 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2025-01-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: COPD; Lung Cancer (NSCLC); Leukemia
Keywords: COPD; Lung cancer; leukemia; Air pollution; Never smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Leukemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Sputum, Exhaled air, Breath condensate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: 150 healthy controls will be recruited as volunteers in the pool of employees of the participating healthcare companies, excluding the participating operational units
- Partecipant: * 50 patients with a histological diagnosis of lung cancer of any histotype and grade according to the World Health Organization (WHO) classification.
  * 50 patients with a diagnosis of COPD according to the ERS/ATS guidelines and GOLD recommendations. The current guidelines define COPD as a chronic lung disease characterized by debilitating symptoms (such as dyspnea, chronic cough with sputum) and caused by exposure to toxic substances such as cigarette smoke and environmental pollutants. The diagnosis is based on the presence of airflow obstruction that is not completely reversible, identified by an FEV1/FVC ratio of <0.7 after bronchodilation testing in subjects with a compatible history.
  * 50 patients with a histological diagnosis of leukemia according to the WHO classification.

SUMMARY:
This study aims to examine the exposure to atmospheric pollutants in a group of non-smoking patients suffering from lung cancer, chronic obstructive pulmonary disease (COPD), and leukemia. The exposure to atmospheric pollutants will be assessed simultaneously in a group of healthy volunteers. The ultimate goal of the study is to enhance the understanding of the mechanisms by which atmospheric pollutants act, in order to develop new tools that can help halt or at least delay the development of diseases associated with pollution.

DETAILED DESCRIPTION:
Atmospheric pollution represents a global issue today. A significant portion of the population in Italy lives in areas where air quality standards are very low, both due to global warming and human-caused pollution. This not only poses a serious risk to human health but also has a tremendous economic and social impact on the National Health System. Atmospheric pollution is associated with a variety of diseases affecting nearly all organs and systems.

In almost all currently available studies on atmospheric pollution and its effects on humans, the population's exposure to pollutants is not measured at the individual level; instead, it is estimated using various environmental sampling techniques based on geographical areas and then applied to individuals based on their residence. There is also a lack of information regarding the effects of confounding risk factors, especially concerning cigarette smoking.

This study aims to acquire more information on the individual exposure to pollutants in a group of non-smoking patients suffering from lung cancer, COPD, and leukemia. The decision to evaluate only never-smokers ensures that there are no confounding factors in the association study between health and environmental pollution.

During a scheduled visit at the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna, the Department of Medical Oncology, IRCCS AOU of Bologna, and the Department of Hematology, Hospital-University Company, Policlinico Riuniti di Foggia, and after obtaining informed consent, the following biological samples will be collected in a non-invasive manner and in small aliquots: exhalate, respiratory condensate, sputum, blood, and urine. The collected samples will then be analyzed by the laboratories of the Occupational Medicine Department (IRCCS - AOU of Bologna) and the Messina Institute of Technology (MeIT) of the Department of Chemical, Biological, Pharmaceutical, and Environmental Sciences (CHIBIOFARAM) of the University of Messina using advanced techniques such as electron microscopy, mass spectrometry chromatography, and for the determination of pollutants such as particulate matter and volatile compounds. Furthermore, the project also aims to identify effect biomarkers involved in the response to such agents.

ELIGIBILITY:
Inclusion Criteria:

Patient Cohort to be Recruited at the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna:

* Age ≥ 18 years
* Patients with a diagnosis of COPD of any severity (FEV1/FVC < 0.7 after bronchodilation test)
* Non-smokers according to ISS definition: patients who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Signature of informed consent

Healthy Volunteer Cohort to be Recruited at the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna:

* Age ≥ 18 years
* Non-smokers according to ISS definition: subjects who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Absence of comorbidities related to the study (COPD, solid tumors, leukemia) in medical history
* Workers of the IRCCS AOU of Bologna, S. Orsola Polyclinic
* Signature of informed consent

Patient Cohort to be Recruited at the Department of Medical Oncology, IRCCS AOU of Bologna:

* Age ≥ 18 years
* Patients with a diagnosis of lung neoplasm of any histotype and stage
* Non-smokers according to ISS definition: patients who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Signature of informed consent

Healthy Volunteer Cohort to be Recruited at the Department of Medical Oncology, IRCCS AOU of Bologna:

* Age ≥ 18 years
* Non-smokers according to ISS definition: subjects who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Absence of comorbidities related to the study (COPD, solid tumors, leukemia) in medical history
* Workers of the IRCCS AOU of Bologna, S. Orsola Polyclinic
* Signature of informed consent

Patient Cohort to be Recruited at the Hematology Department (Hospital-University Company, Policlinico Riuniti di Foggia):

* Age ≥ 18 years
* Non-smokers according to ISS definition: patients who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Patients with a diagnosis of leukemia of any type
* Signature of informed consent

Healthy Volunteer Cohort to be Recruited at the Hematology Department (Hospital-University Company, Policlinico Riuniti di Foggia):

* Age ≥ 18 years
* Non-smokers according to ISS definition: subjects who declare having smoked less than 100 cigarettes (5 packs of 20) in their lifetime and are not currently smokers
* Absence of comorbidities related to the study (COPD, solid tumors, leukemia) in medical history
* Workers of the Hospital-University Company, Policlinico Riuniti di Foggia
* Signature of informed consent

Exclusion Criteria:

Patient Cohort to be Recruited at the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna:

* Deficiency of alpha-1 antitrypsin (A1AT)

Healthy Volunteer Cohort to be Recruited at the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna:

* Workers from the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna, S. Orsola Polyclinic

Patient Cohort to be Recruited at the Department of Medical Oncology, IRCCS AOU of Bologna:

* Previous and/or current diagnosis of solid tumors, myelodysplastic syndromes, myeloproliferative neoplasms
* Previous and/or current treatment with antineoplastic agents

Healthy Volunteer Cohort to be Recruited at the Department of Medical Oncology, IRCCS AOU of Bologna:

* Workers from the Department of Medical Oncology, IRCCS AOU of Bologna, S. Orsola Polyclinic

Patient Cohort to be Recruited at the Hematology Department (Hospital-University Company, Policlinico Riuniti di Foggia):

* Previous diagnosis of solid tumors, myelodysplastic syndromes, myeloproliferative neoplasms
* Previous treatment with antineoplastic agents (alkylating agents, hydroxyurea, topoisomerase II inhibitors, lenalidomide) -Presence of pre-existing genetic conditions (Fanconi anemia, ataxia- telangiectasia, Down syndrome, xeroderma pigmentosum, Li-Fraumeni syndrome)
* Infection with human immunodeficiency virus (HIV), human T-lymphotropic virus types 1 or 2, or Epstein-Barr virus

Healthy Volunteer Cohort to be Recruited at the Hematology Department (Hospital-University Company, Policlinico Riuniti di Foggia):

* Workers from the Hematology Department, Hospital-University Company, Policlinico Riuniti di Foggia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients affected by COPD, lung cancer, and leukemia, attending the Department of Pneumology and Respiratory Intensive Care, IRCCS AOU of Bologna, the Department of Medical Oncology, IRCCS AOU of Bologna, and the Hematology Department, Hospital-University Company, Policlinico Riuniti di Foggia.
  Healthy controls will also be recruited as volunteers from the pool of employees of the participating healthcare facilities, excluding the participating operating units.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Scanning Electron Microscopy (SEM): presence of inorganic and organic particulate matter
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Transmission Electron Microscopy (TEM): presence of inorganic and organic particulate matter
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Atomic Force Microscopy (AFM): presence of inorganic and organic particulate matter
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Infrared (IR) and Raman Spectroscopy: presence of inorganic and organic particulate matter
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Inductively Coupled Plasma Mass Spectrometry (ICP-MS): presence of metals
Identification of pollutants in biological samples | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months."
  -Gas Chromatography-Mass Spectrometry (GC-MS): presence of volatile compounds (e.g., VOCs) and semi-volatile compounds

SECONDARY OUTCOMES:
Evaluation of the association between the identified pollutants and the development of COPD, lung cancer, and leukemia in a population of patients who have never smoked. | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months.
  The objective will be measured by comparing the concentration (units/volume) of the identified pollutants within the biological samples of patients affected by lung cancer, COPD, and leukemia with those identified in the biological samples of healthy subjects, collected through:
  * Scanning Electron Microscopy (SEM): presence of inorganic and organic -particulate matter
  * Transmission Electron Microscopy (TEM): presence of inorganic and organic particulate matter
  * Atomic Force Microscopy (AFM): presence of inorganic and organic particulate matter
  * Infrared (IR) and Raman Spectroscopy: presence of inorganic and organic particulate matter
  * Inductively Coupled Plasma Mass Spectrometry (ICP-MS): presence of metals Gas Chromatography-Mass Spectrometry (GC-MS): presence of volatile compounds (e.g., VOCs) and semi-volatile compounds
Identification of potential effect biomarkers involved in the response to pollutants. | The collection of biological samples will be conducted during the enrollment visit, and the analyses will be carried out over the following 18 months
  The objective will be measured by evaluating the alteration of endogenous molecule content (biomarkers) in the presence of the identified pollutants through the conduction of dose-response curves.
  High-Performance Liquid Chromatography/Mass Spectrometry (HPLC-MS) Gas Chromatography-Mass Spectrometry (GC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - Medical Oncology, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Respiratory and Critical Care Unit, IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bologna
  - Ematology Unit, Azienda Ospedaliero-Universitaria, Policlinico Riuniti di Foggia, Foggia, Foggia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun Q, Wang B, Xu S, Cong X, Pu Y, Zhang J. Research development and trends of benzene-induced leukemia from 1990 to 2019-A bibliometric analysis. Environ Sci Pollut Res Int. 2022 Feb;29(7):9626-9639. doi: 10.1007/s11356-021-17432-3. Epub 2022 Jan 8. PMID 34997503
- [Result] Wang X, Chen L, Cai M, Tian F, Zou H, Qian ZM, Zhang Z, Li H, Wang C, Howard SW, Peng Y, Zhang L, Bingheim E, Lin H, Zou Y. Air pollution associated with incidence and progression trajectory of chronic lung diseases: a population-based cohort study. Thorax. 2023 Jul;78(7):698-705. doi: 10.1136/thorax-2022-219489. Epub 2023 Feb 2. PMID 36732083